CLINICAL TRIAL: NCT02880254
Title: A Study to Assess the Compliance and Impact on Weight of Kurbo, a Pediatric Centered Weight Loss App
Acronym: Kurbo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Rushika Conroy, Assistant Professor of Pediatrics, Tufts University School of Medicine, Baystate Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 891748
Record Dates: First submitted 2016-08-15; First posted 2016-08-26 (Estimated); Results first posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Obesity
Keywords: body mass index change; weight loss; patient compliance
MeSH Terms: conditions — Obesity; Weight Loss; Patient Compliance

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kurbo only (Active Comparator): use of app plus standard of care
  Interventions: Device: Kurbo
- Kurbo plus PHC (Active Comparator): use of app, personal health coach and standard of care
  Interventions: Device: Kurbo; Device: Personal Health Coach

INTERVENTIONS:
Device: Kurbo — health/weight loss app designed for children and adolescents to help them track intake, output and understand healthy eating habits
Device: Personal Health Coach — weekly health coach via facetime or Skype to motivate and counsel subjects during the weight loss process
  Arms: Kurbo plus PHC

SUMMARY:
Kurbo is a health and fitness app that is targeted toward the pediatric population. It utilizes games and activities to educate children about healthy eating, portion control/size and exercise. It allows for food tracking by using servings of macronutrients and food groups and sets goals for achieving a healthy BMI through modification of diet intake. In addition to being created solely for children and adolescents, a unique feature of this app is an option to speak with a personal health coach on a regular basis to obtain feedback, advice and encouragement. Studies suggest that weight loss outcomes are best with more frequent contact hours but most weight loss clinics, including ours, are not equipped to meet with patients on a weekly basis or even monthly basis. The personal coaching aspect of Kurbo is expected to improve outcomes by increasing user access to feedback and advice.

The purpose of this pilot study is to assess the feasibility, compliance with and effects of a pediatric centered weight loss app on BMI z-scores in a group of children and adolescents in a pediatric weight management program. The investigators will assess the impact of the app as an adjunct to current weight management therapy, both with and without the personal health coach (PHC) option.

DETAILED DESCRIPTION:
As a result of childhood obesity and its comorbidities, this generation of children might be the first to not outlive its parents. The national prevalence of adolescent obesity has increased from 5% to 21% over the last five decades. Even more discouraging is that youth are being afflicted with the same obesity-related comorbidities that are affecting adults. Conditions such as type 2 diabetes, hypertension, non-alcoholic fatty liver disease, dyslipidemia, metabolic syndrome, and sleep apnea are being diagnosed in children at younger and younger ages.

Lifestyle modification continues to be the cornerstone of treatment for obesity and its associated conditions. The basic concept behind lifestyle modification is a balance of caloric intake and caloric output. Lifestyle modification alone has shown to result in on average 5-10% weight loss over a 6 month period in adults or a 1-2 kg weight loss over 6-12 months. In pediatrics, weight loss is generally not used a marker of success given that the child is still growing linearly in most cases. Thus, changes in BMI and/or BMI z-score are utilized to measure success. Pediatric studies cite improvements in BMI z-score ranging from 0.004 to 0.42 with most studies averaging a 0.1-0.2 decrease in BMI z- score over 6 to 12 months.

The pediatric weight management program at Baystate Medical Center sees children and adolescents from the ages of 2-20 years. Standard care for the program involves monthly visits with a physician (either a general pediatrician or pediatric endocrinologist) or a nurse practitioner in addition to visits every 3 months with a registered dietitian. During each visit, food and activity recalls are conducted and 1-2 goals are made with the patient and their caregivers that focus on improving the quality and quantity of the patient's intake as well as increasing physical activity. Goals are personalized and are adjusted to meet the social, psychological, financial and motivational needs of the patient.

Sixty four percent of Americans own smartphones. The use of smartphone apps for health and wellness has sky rocketed as more sophisticated and user friendly apps are being developed to assist with weight loss, healthy eating, exercise and tracking food and activity. Digital tools can allow one to be constantly aware of how much they are eating and expending, which may result in an improvement in overall weight loss. In adults weight loss of 1-5 kg over a 6 month period is achievable using tools such as food log apps. Such apps are generally suited for adults only and the few weight loss apps targeted toward the pediatric population have not been validated by weight loss programs. Apps that are available for younger patients have been criticized for containing inadequate expert recommended strategies for achieving a healthy weight, lack of goal setting, and poor provision of education.

Kurbo is a health and fitness app that is targeted toward the pediatric population. It utilizes games and activities to educate children about healthy eating, portion control/size and exercise. It allows for food tracking by using servings of macronutrients and food groups and sets goals for achieving a healthy BMI through modification of diet intake. In addition to being created solely for children and adolescents, a unique feature of this app is an option to speak with a personal health coach on a regular basis to obtain feedback, advice and encouragement. Studies suggest that weight loss outcomes are best with more frequent contact hours but most weight loss clinics, including ours, are not equipped to meet with patients on a weekly basis or even monthly basis. The personal coaching aspect of Kurbo is expected to improve outcomes by increasing user access to feedback and advice.

The purpose of this pilot study is to assess the feasibility, compliance with and effects of a pediatric centered weight loss app on BMI z-scores in a group of children and adolescents in a pediatric weight management program. The investigators will assess the impact of the app as an adjunct to current weight management therapy, both with and without the personal health coach (PHC) option.

The Primary aim is to assess 3 month compliance with the Kurbo app as well as the Kurbo app and PHC by a group of morbidly obese children and adolescents in a weight management program. The investigators hypothesize that compliance with the Kurbo app and Kurbo app plus PHC will be better than known compliance of the investigators standard of care group. The Secondary aim is to assess the effect of the Kurbo app as well as the Kurbo app and PHC on 3 month change in BMI-z score among morbidly obese children and adolescents undergoing a weight management program. The hypothesis is that the use of the Kurbo app and Kurbo app plus a personal health coach will result in a greater reduction in BMI z-score over 3 months than known change in a standard care group and that the use of the app and personal health coach will result in a greater reduction in BMI z-score over 3 months than with the use of the app without the personal health coach.

ELIGIBILITY:
Inclusion Criteria:

1. At least 10 years and no more than 17 years of age
2. New patients presenting to the Baystate Children's Hospital pediatric weight management program

Exclusion Criteria:

1. Do not own or have regular access to a smartphone
2. Cannot read and understand English language as Kurbo is currently only designed for English speakers

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2016-09; Primary Completion 2018-01-01 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rushika Conroy, MD MS, Principal Investigator — Baystate Medical Center

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available within 1 year of study completion.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Booth HP, Prevost TA, Wright AJ, Gulliford MC. Effectiveness of behavioural weight loss interventions delivered in a primary care setting: a systematic review and meta-analysis. Fam Pract. 2014 Dec;31(6):643-53. doi: 10.1093/fampra/cmu064. Epub 2014 Oct 8. PMID 25298510
- [Background] Muhlig Y, Wabitsch M, Moss A, Hebebrand J. Weight loss in children and adolescents. Dtsch Arztebl Int. 2014 Nov 28;111(48):818-24. doi: 10.3238/arztebl.2014.0818. PMID 25512008
- [Background] Cheng JK, Wen X, Coletti KD, Cox JE, Taveras EM. 2-Year BMI Changes of Children Referred for Multidisciplinary Weight Management. Int J Pediatr. 2014;2014:152586. doi: 10.1155/2014/152586. Epub 2014 Jan 30. PMID 24672556
- [Background] Carter MC, Burley VJ, Nykjaer C, Cade JE. Adherence to a smartphone application for weight loss compared to website and paper diary: pilot randomized controlled trial. J Med Internet Res. 2013 Apr 15;15(4):e32. doi: 10.2196/jmir.2283. PMID 23587561
- [Background] Flores Mateo G, Granado-Font E, Ferre-Grau C, Montana-Carreras X. Mobile Phone Apps to Promote Weight Loss and Increase Physical Activity: A Systematic Review and Meta-Analysis. J Med Internet Res. 2015 Nov 10;17(11):e253. doi: 10.2196/jmir.4836. PMID 26554314
- [Background] Franz MJ, VanWormer JJ, Crain AL, Boucher JL, Histon T, Caplan W, Bowman JD, Pronk NP. Weight-loss outcomes: a systematic review and meta-analysis of weight-loss clinical trials with a minimum 1-year follow-up. J Am Diet Assoc. 2007 Oct;107(10):1755-67. doi: 10.1016/j.jada.2007.07.017. PMID 17904936
- See also: 5. Pew Research Center, April, 2015, "The Smartphone Difference" — http://www.pewinternet.org/2015/04/01/us-smartphone-use-in-2015

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: difficulty recruiting participants to be in the trial in the time frame; some agreed but then never came in to consent; there were no patients who consented but did not participate
Period: Overall Study
Arm/Group | Kurbo Only | Kurbo Plus PHC
Started | 13 | 14
Completed | 4 | 4
Not Completed | 9 | 10

BASELINE CHARACTERISTICS:
Population: We had no patients who consented but did not participate in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Kurbo Only | Kurbo Plus PHC | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 14 | 27
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.1 (2) | 13 (2.9) | 13 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: 3 Month Compliance With the Kurbo App as Well as the Kurbo App and PHC by a Group of Morbidly Obese Children and Adolescents in a Weight Management Program.
Description: A questionnaire will be handed out to each subject every month (see below) where applicable.we will utilize one-sample tests with a one-sided alpha of 0.025. One-sided tests will be used as we are only interested in whether the use of this app results in better outcomes than usual care. Compliance will utilize a binomial probability test to assess compliance against our known compliance of 50%.
  Questionnaire is noted here:
  Confidential Page 1 of 1 Kurbo Survey [baseline_arm_1][name], DOB [baseline_arm_1][dob] Please complete the survey below. Thank you! Group Allocation __________________________________ Who is completing this survey? Child / Patient Parent / Guardian Over the last month, abou
Time Frame: 3 months
Population: Assuming we find improved compliance and BMI-z scores, we will estimate compliance and BMI-z score differences between Kurbo and Kurbo + PHC. Estimates will be generated using direct observation as well as prediction through modeling.
Measure: Number; unit: percent compliant
Arm/Group | Kurbo Only | Kurbo Plus PHC
Number analyzed (Participants) | 13 | 14
percent compliant
  compliance with food tracking | 0 | 14
  compliance with exercise tracking | 0 | 7

2. Secondary Outcome: the Effect of the Kurbo App as Well as the Kurbo App and PHC on 3 Month Change in BMI Zscore Among Morbidly Obese Children and Adolescents Undergoing a Weight Management Program.
Description: BMI zscore will be determined from mathematical calculations derived from subject's height and weight. Z score is the number of standard deviations from the mean. A Z score of 0 is the mean. A change in z score in the positive direction reflects an increase in BMI Z score. A change in z score in the negative direction reflects a decrease in BMI Z score. A decrease in BMI z score indicates a change in BMI that favors weight loss.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: z score
Arm/Group | Kurbo Only | Kurbo Plus PHC
Number analyzed (Participants) | 13 | 14
z score | 2.4 (0.3) | 2.2 (0.3)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Kurbo Only | Kurbo Plus PHC
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/54/NCT02880254/Prot_SAP_000.pdf